CLINICAL TRIAL: NCT07210060
Title: Comparison of Knee Strengthening Combined With Hip or Ankle Joint Exercises on Clinical Symptoms, Sports Performance and Soft Tissue Structure in Women With Patellofemoral Pain Syndrome
Brief Title: Knee Strengthening With Hip vs. Ankle Exercises in Women With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-E(I)-20220334
Record Dates: First submitted 2025-09-18; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain; Exercise Therapy
Keywords: Dynamic alignment; Tele-rehabilitation; Pain modulation; Muscle strength
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Papaverine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HK group (Experimental): hip + knee joint exercise group
  Interventions: Other: hip + knee joint exercise group
- AK group (Experimental): ankle + knee joint exercise group
  Interventions: Other: ankle + knee joint exercise group
- Stretching group (Sham Comparator): Stretching group
  Interventions: Other: Stretching group

INTERVENTIONS:
Other: hip + knee joint exercise group — Hip: squat, glute bridge and gluteus medius exercise Knee: knee flexor and extensor, isometric squat hold
  Arms: HK group
Other: ankle + knee joint exercise group — Knee: knee flexor and extensor, isometric squat hold Ankle: plantar flexor, dorsi flexor and lunge
  Arms: AK group
Other: Stretching group — Education Handout on Lower Limb Stretching
  Arms: Stretching group

SUMMARY:
Eight weeks of telehealth-based supervised exercise effectively reduced DKV and pain in women with anterior knee pain. Both intervention groups demonstrated comparable benefits.

DETAILED DESCRIPTION:
This study compared the effects of knee strengthening combined with either hip or ankle joint exercises on dynamic knee valgus (DKV), visual analogue scale (VAS) scores during activity, tendon stiffness, muscle structure, ankle range of motion, and muscle strength in women with anterior knee pain. Forty-five female recreational athletes aged 20-40 with anterior knee pain were randomly assigned to three groups: hip + knee exercises (HK group, n = 15), ankle + knee exercises (AK group, n = 15), and stretching alone (control group, n = 15). The HK and AK groups received supervised telehealth-based exercise sessions (30 minutes/day, 3 times/week for 8 weeks), while the control group received only an educational pamphlet. Assessments were conducted at baseline, 4 weeks, and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Female recreational athletes aged 20-40 years who engage in regular exercise
2. Experiencing pain in the anterior or surrounding patella during at least two or more of the following activities: walking, running, jumping, kneeling, squatting, climbing stairs, or prolonged sitting
3. A pain index of 3 or higher on the Numeric Pain Rating Scale (NPRS) and symptoms persisting for at least 3 months
4. Knee pain unrelated to trauma.

Exclusion Criteria:

1. Inability to operate a smartphone or computer
2. History of fractures or surgeries involving the hip, knee, ankle, or foot
3. History of meniscus, knee ligament injuries, or ankle sprains within the last six months
4. Knee ligament laxity, inflammation, swelling, patellar dislocation, or subluxation
5. Cognitive impairment or inability to follow simple instructions
6. History of cardiovascular or neurological disorders
7. Advised by a physician to avoid exercise. Use of over-the-counter pain medication was not an exclusion criterion.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Single Leg Landing Task | 2 minute
  The participant stood on a 30 cm box and first bent the non-testing leg's knee to approximately 90 degrees. After stabilizing, the participant jumped forward with the testing leg to a target 10 cm away from the box, maintaining balance for five seconds upon landing.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 1 minute
  0 indicates no pain and 10 indicates the worst pain imaginable.
Patellar Tendon Stiffness Measurement | 3 minute
  The stiffness of the patellar tendon was assessed using a handheld device (MyotonPRO; Tallinn, Estonia).
Muscle structure | 15 minute
  A portable ultrasound device (Linear wireless probe LU700L VET) was used to assess the structure of the gastrocnemius and gluteus medius muscles in a resting state.
Ankle Joint ROM | 3 minute
  used a weight-bearing lunge test to measure the active dorsiflexion angle of the ankle during weight-bearing.
Maximum Voluntary Isometric Strength | 15 minute
  A handheld dynamometer (MicroFET3; Hoggan Scientific LLC, USA) was used to measure the maximum isometric strength of the hip abductors, knee extensors, ankle dorsiflexors, and ankle plantar flexors.

CONTACTS AND LOCATIONS:
Locations (1):
- Nai-Jen Chang, Tainan, Kaohsiung City, Taiwan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT07210060/Prot_SAP_000.pdf